CLINICAL TRIAL: NCT00194532
Title: Cefpodoxime vs Ciprofloxacin for Acute Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27085-D
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2011-04-28 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Urinary Tract Infection
Keywords: UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cefpodoxime; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefpodoxime (Experimental): Cefpodoxime 100mg twice a day(BID)for 3 days
  Interventions: Drug: Cefpodoxime
- Ciprofloxacin (Active Comparator): Ciprofloxacin 250mg twice a day (BID)for 3 days
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Cefpodoxime — Cefpodoxime 100mg twice a day(BID)for 3 days
  Arms: Cefpodoxime
Drug: Ciprofloxacin — Ciprofloxacin 250mg twice a day (BID)for 3 days
  Arms: Ciprofloxacin

SUMMARY:
Urinary tract infection (UTI) is a very common problem in young healthy women, afflicting approximately one-half of women by their late 20s. One of the most common antibiotics used to treat UTIs is ciprofloxacin, usually for a total of three days. However, increasing resistance to this antibiotic has raised concerns about its overuse for cystitis and generated interest in alternative agents. An alternative antibiotic which is approved for use in UTIs is cefpodoxime. However, there are few studies evaluating the efficacy and tolerance of this compound when given in a 3-day regimen as is commonly used for treatment of UTI. The major purpose of this study is to assess the efficacy and tolerance of a 3-day regimen of cefpodoxime versus ciprofloxacin for treatment of acute uncomplicated cystitis.

DETAILED DESCRIPTION:
Procedures subjects will undergo once they have read and signed the consent are:

Questions about their medical and sexual history and current symptoms of UTI. They will be asked to provide a urine and peri-urethral sample and then are randomly assigned to one of the two treatment groups.They will be given a sheet to record symptoms at home. They will be asked to return to the clinic in 5-9 and 28-30 days after completing antibiotic therapy.Follow-up questions will be asked and urine and peri-urethral will be self collected at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant females in good general health with symptoms of acute cystitis

Exclusion Criteria:

* Pregnant,lactating, or not regularly contracepting: known anatomic abnormalities of the urinary tract; use of prophylactic antibiotics; history of allergy or intolerance to any of the study drugs; recent (>2 weeks)exposure to an oral or parenteral antimicrobial; or history of UTI in the previous 1 month

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2005-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Stapleton, MD, Principal Investigator — University of Washington, Department of Medicine
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Hooton TM, Roberts PL, Stapleton AE. Cefpodoxime vs ciprofloxacin for short-course treatment of acute uncomplicated cystitis: a randomized trial. JAMA. 2012 Feb 8;307(6):583-9. doi: 10.1001/jama.2012.80. PMID 22318279

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin: Ciprofloxacin 250 mg BID X 3 days
- Cefpodoxime: Cefpodoxime 100 mg BID X 3 days
Period: Overall Study
Arm/Group | Ciprofloxacin | Cefpodoxime
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Cefpodoxime | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Full Range); unit: years] | 24 [18 to 55] | 23 [17 to 44] | 24 [17 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 150 | 300
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure
Description: Participants with clinical cure, i.e. free of urinary tract symptoms and requiring no further antibiotic treatment, to assess the efficacy of a 3-day regimen of cefpodoxime compared to ciprofloxacin
Time Frame: 28-30 days post therapy
Population: modified ITT
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin | Cefpodoxime
Number analyzed (Participants) | 150 | 150
participants
  Cure | 140 | 123
  Not cure | 10 | 27

2. Secondary Outcome: Microbiologic Cure
Description: Elimination or decrease of causative uropathogen(s) in the mid-stream urine culture at follow-up
Time Frame: 1-15 days post therapy
Population: Per protocol. Participants were eligible for analysis if they had an enrollment urine containing uropathogens and a urine specimen taken at follow-up.
Measure: Number; unit: participants
Arm/Group | Ciprofloxacin | Cefpodoxime
Number analyzed (Participants) | 128 | 129
participants
  Cure | 123 | 104
  Not cure | 5 | 25

ADVERSE EVENTS:
Arm/Group | Ciprofloxacin | Cefpodoxime
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 41/137 | 37/137
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin (N=137) | Cefpodoxime (N=137)
gastrointestinal(GI) side effects (Gastrointestinal disorders) | 23 (30) | 21 (26) — nausea, vomiting, loose stools, abdominal discomfort, other GI
central nervous system (CNS) side effect (Nervous system disorders) | 17 (18) | 15 (16) — headache, dizziness
vaginal side effects (Reproductive system and breast disorders) | 8 (8) | 7 (7) — vaginal discomfort, discharge, itching, or self-diagnosed yeast
nausea (Gastrointestinal disorders) | 13 (13) | 8 (8) — included under GI side effects
loose stools (Gastrointestinal disorders) | 7 (7) | 9 (9) — included under GI side effects
abdominal discomfort (Gastrointestinal disorders) | 7 (7) | 7 (7) — included under GI side effects
headache (Nervous system disorders) | 4 (4) | 7 (7) — included under CNS side effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes